CLINICAL TRIAL: NCT02483780
Title: Culturally Adaptive Storytelling Method to Improve Hypertension Control in Vietnam -"We Talk About Our Hypertension": a Pilot Cluster Randomized Controlled Trial
Brief Title: We Talk About Our Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Population, Health and Development, Vietnam (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014/PHAD/UMMS 01-01
Record Dates: First submitted 2015-06-22; First posted 2015-06-29 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Storytelling intervention (Experimental): Two communes will be assigned to intervention group. Within each commune, 25 adults with HTN will be enrolled.
  Patients will receive 2 DVDs with stories of patients who have successfully controlled their hypertension and "Learn More" section, which will be coordinated with specific patient stories and will fill in gaps not covered by the storytellers.
  Interventions: Behavioral: Storytelling
- Usual care (No Intervention): Two communes will be assigned to usual care group. Within each commune, 25 adults with HTN will be enrolled.
  Patients will receive 2 DVDs with only didactic material about common non-communicable diseases but without hypertension related stories.

INTERVENTIONS:
Behavioral: Storytelling — The intervention will center on stories about living with hypertension, with patients speaking in their own words.
  Arms: Storytelling intervention

SUMMARY:
The proposed pilot community-based research project will examine the feasibility, acceptability, and potential efficacy of the Storytelling intervention compared with usual care in hypertension control among rural residents in 4 communities in Vietnam. This is a major clinical and public health problem in this developing country.

ELIGIBILITY:
Inclusion Criteria:

Consenting adult men and women must fulfill each of the following criteria:

1. be a resident of the selected commune;
2. be aged 50 years or older;
3. have a diagnosis of hypertension according to the 7th Joint National Commission of High Blood Pressure (JNC 7)
4. not be cognitively impaired (as assessed by study physicians)
5. not be a "story teller" used to develop the intervention;
6. not be a family member of another participant in the study

Exclusion Criteria:

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
recruitment rate | 3 months
retention rate | 1 year

SECONDARY OUTCOMES:
Blood pressure | 3 months after randomization
  systolic and diastolic BP and the proportion of participants with controlled BP defined as in JNC-8

CONTACTS AND LOCATIONS:
Overall Officials: Hoa Nguyen, MD, Ph.D, Study Director — Institute of Population, Health and Development
Locations (1):
- Institute of Population, Health and Development (PHAD), Hà Nội, Vietnam

REFERENCES:
- [Derived] Nguyen HL, Ha DA, Goldberg RJ, Kiefe CI, Chiriboga G, Ly HN, Nguyen CK, Phan NT, Vu NC, Nguyen QP, Allison JJ. Culturally adaptive storytelling intervention versus didactic intervention to improve hypertension control in Vietnam- 12 month follow up results: A cluster randomized controlled feasibility trial. PLoS One. 2018 Dec 31;13(12):e0209912. doi: 10.1371/journal.pone.0209912. eCollection 2018. PMID 30596749
- [Derived] Nguyen HL, Allison JJ, Ha DA, Chiriboga G, Ly HN, Tran HT, Nguyen CK, Dang DM, Phan NT, Vu NC, Nguyen QP, Goldberg RJ. Culturally adaptive storytelling intervention versus didactic intervention to improve hypertension control in Vietnam: a cluster-randomized controlled feasibility trial. Pilot Feasibility Stud. 2017 May 1;3:22. doi: 10.1186/s40814-017-0136-9. eCollection 2017. PMID 28473924
- [Derived] Allison JJ, Nguyen HL, Ha DA, Chiriboga G, Ly HN, Tran HT, Phan NT, Vu NC, Kim M, Goldberg RJ. Culturally adaptive storytelling method to improve hypertension control in Vietnam - "We talk about our hypertension": study protocol for a feasibility cluster-randomized controlled trial. Trials. 2016 Jan 14;17:26. doi: 10.1186/s13063-015-1147-6. PMID 26762128